CLINICAL TRIAL: NCT05677399
Title: The Effectiveness of Peloidotherapy and Aquatic Exercise in Knee Osteoarthritis Treatment.
Brief Title: Knee Osteoarthritis Treatment With Peloidotherapy and Aquatic Exercise.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Arel University (Other)
Responsible Party: Principal Investigator, Seçil ÖZKURT, Asst. Prof. Dr., Istanbul Arel University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5000007
Record Dates: First submitted 2023-01-03; First posted 2023-01-10 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Knee Osteoarthritis
Keywords: knee osteoarthritis; peloidotherapy; aquatic exercise; water based exercise; balneotherapy; aquatic rehabilitation
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: A Randomized, single blind, prospective, parallel 1:1 group study.
Who Masked: Outcomes Assessor
Masking Description: Patients were assessed before treatment, after treatment, 1 month after treatment and 3 month after treatment by the investigator (İ.T.) who was blinded to the study. İ.T. is medical doctor who didn't know the patients' groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): Treatment group received 30 minutes of aquatic exercise by a physiotherapist in a warmed up to 33° C tap water and 30 minutes of mud pack treatment at 42°C on both knees 5 weekdays for 2 consecutive weeks (totally 10 sessions).
  Interventions: Other: aquatic exercise and peloidotherapy
- Control Group (No Intervention): Control group continued to use their usual medical treatment.

INTERVENTIONS:
Other: aquatic exercise and peloidotherapy — Treatment group received 30 minutes of aquatic exercise by a physiotherapist in a warmed up to 33° C tap water and 30 minutes of mud pack treatment at 42°C on both knees 5 weekdays for 2 consecutive weeks (totally 10 sessions).
  Other Names: water based exercise and mud pack therapy
  Arms: Treatment Group

SUMMARY:
The aim was to observe the short and medium term effects of peloidotherapy and aquatic exercise applications in patients with knee osteoarthritis.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is one of the most common musculoskeletal diseases in the world. It is a non-inflammatory chronic disease that starts from the articular cartilage and is characterized by mechanical wear and cartilage loss in the joints, and includes findings such as joint pain, stiffness, and limitation of movement. Its incidence increases with aging. OA is more common in the spine, hip, hand and knee joints. The knee, which is a load-bearing joint, is more affected. Knee osteoarthritis is one of the most common causes of disability. It is more common in women. The prevalence of symptomatic knee osteoarthritis in adults over the age of 55 was found to be 13% In the treatment guidelines, aquatic exercise and balneotherapy are among the recommendations for knee OA. Balneotherapy is a stimulus performed at a certain time interval and in a cure style, by using thermal and/or mineral waters, peloids (medical mud) and gases, in the form of bath, package, drinking and inhalation applications, whose methods and doses have been determined. compliance therapy. There are clinical studies showing that balneotherapy and mud pack applications reduce pain and increase functional capacity in knee osteoarthritis. Odabaşı et al. showed that peloidotherapy, one of the balneological methods, has not only thermic effect but also chemical effect in the treatment of knee OA. In patients with knee OA, pain, physical disability, quadriceps femoris muscle weakness and limitations in joint range of motion are observed. it reduces the level of physical activity, exercise capacity and quality of life in these people. The fact that the body is supported due to the buoyancy of the water in the exercises performed in the water reduces the load on the joints during the movement. For this reason, many movements that cannot be done on land can be done safely in water. On the other hand, because the density of water is higher than air, the muscles have to do more work even when performing a simple movement in water compared to the movements on land. Special rehabilitation programs based on water exercise programs have started to be one of the applications that can be done to increase muscle strength for these reasons.

When the literature was reviewed, we could not find any study examining the combination of aquatic exercise and peloid application in patients with knee osteoarthritis.

The aim of this study was to evaluate the effects of co-administration of peloid and aquatic exercises in knee osteoarthritis patients with a single-blind randomized controlled study.

ELIGIBILITY:
Inclusion Criteria:

* primary knee osteoarthritis diagnosed according to the ACR criteria
* gave their written informed consent
* 40-75 ages
* Kellgren Lawrence grading 2-4
* having symptomatic knee pain at least 3 months.

Exclusion Criteria:

* secondary knee OA
* pathology of the waist, hip, or ankle joints
* decompensated organ failure
* malignancy,
* active bleeding
* infectious disease
* serious knee injuries or previous surgical procedures within the past 6 months
* the use of intraarticular steroids and hyaluronic acid injection to the knee joint within the past 6 months
* physiotherapy, balneotherapy, or peloidotherapy within the past 1 year.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2015-09-09 (Actual); Primary Completion 2016-06-10 (Actual); Study Completion 2016-12-10 (Actual)

PRIMARY OUTCOMES:
Pain (VAS) | Change from baseline pain (VAS) at the end of the treatment, 1 month after treatment ,3 months after treatment.
  The VAS is a commonly used scale which determines the intensity of pain. It consists of a 10-cm long line, drawn horizontally Numeric value (in cm between 0 and 10) of patients' pain intensity was determined by measuring the distance between the lowest VAS value and patients' marks.
WOMAC (total) | Change from baseline WOMAC scores at the end of the treatment, 1 month after treatment ,3 months after treatment.
  The WOMAC Scale is a commonly used well-being scale for patients with knee or hip OA. It consists of three main sections: pain, stiffness, and physical function. It contains a total of 24 items. Scoring of these items is done according to the Likert scale. In the Likert scale, patients indicate pain and difficulty levels by giving scores between 0 and 4. Turkish validity and reliability study had been conducted for WOMAC

SECONDARY OUTCOMES:
IGA (VAS) | Change from baseline IGA (VAS) at the end of the treatment, 1 month after treatment ,3 months after treatment.
  Investivagors' Global Assessment. The VAS is a commonly used scale which determines the intensity of pain. It consists of a 10-cm long line, drawn horizontally Numeric value (in cm between 0 and 10) of patients' pain intensity was determined by measuring the distance between the lowest VAS value and patients' marks.Also is used to assess the patients' global and physicians' global assessment.
PGA (VAS) | Change from baseline PGA (VAS) at the end of the treatment, 1 month after treatment ,3 months after treatment.
  Patients' Global Assessment. The VAS is a commonly used scale which determines the intensity of pain. It consists of a 10-cm long line, drawn horizontally Numeric value (in cm between 0 and 10) of patients' pain intensity was determined by measuring the distance between the lowest VAS value and patients' marks.Also is used to assess the patients' global and physicians' global assessment.
WOMAC (pain) | Change from baseline WOMAC (pain) scores at the end of the treatment, 1 month after treatment ,3 months after treatment.
  The WOMAC Scale is a commonly used well-being scale for patients with knee or hip OA. It consists of three main sections: pain, stiffness, and physical function. It contains a total of 24 items. Scoring of these items is done according to the Likert scale. In the Likert scale, patients indicate pain and difficulty levels by giving scores between 0 and 4. Turkish validity and reliability study had been conducted for WOMAC.
WOMAC (stiffness) | Change from baseline WOMAC (stiffness) scores at the end of the treatment, 1 month after treatment ,3 months after treatment.
  The WOMAC Scale is a commonly used well-being scale for patients with knee or hip OA. It consists of three main sections: pain, stiffness, and physical function. It contains a total of 24 items. Scoring of these items is done according to the Likert scale. In the Likert scale, patients indicate pain and difficulty levels by giving scores between 0 and 4. Turkish validity and reliability study had been conducted for WOMAC.
WOMAC (physical function) | Change from baseline WOMAC (physical function) at the end of the treatment, 1 month after treatment ,3 months after treatment.
  The WOMAC Scale is a commonly used well-being scale for patients with knee or hip OA. It consists of three main sections: pain, stiffness, and physical function. It contains a total of 24 items. Scoring of these items is done according to the Likert scale. In the Likert scale, patients indicate pain and difficulty levels by giving scores between 0 and 4. Turkish validity and reliability study had been conducted for WOMAC.
LAFI | Change from baseline LAFI at the end of the treatment, 1 month after treatment ,3 months after treatment.
  LAFI is used to determine the pain and functional severity of knee and hip OA with three parts of pain, maximum walk distance and some activities of daily living. It has 11 questions of total score of 0 to 24 that higher scores shows more involvement
HAQ | Change from baseline HAQ at the end of the treatment, 1 month after treatment ,3 months after treatment.
  HAQ is used to evaluate functional disability status of patients in eight subscales; dressing, rising, eating, walking, hygiene, reach, grip and usual activities. It includes 20 items and each item has 3 likert score which 0 to 3 where 3 is unable to do
SF-36 | Change from baseline SF-36 at the end of the treatment, 1 month after treatment ,3 months after treatment.
  The SF-36 Health Survey is a comprehensive measurement tool used to evaluate non-disease-specific overall quality of life. It has been developed and made available by Rand Corporation in order to evaluate overall quality of life (). It contains a total of 36 items with eight subscales: physical functioning, role-physical, role-emotional, bodily pain, social functioning, mental health, vitality, and general health. It grades the patient by using scores between 0 and 100,0 indicating poor health while 100 indicating good health. Turkish validity and reliability study had been con¬ducted for SF-36
Timed Up and Go Test | Change from baseline TUG at the end of the treatment, 1 month after treatment ,3 months after treatment.
  TUG is a valid and reliable functional mobility test. It has a correlation with lower extremity strength and useful for identifying older adults risk of falling